CLINICAL TRIAL: NCT03317535
Title: Choice of Anesthesia for Endovascular Treatment of Acute Ischemic Stroke in Posterior Circulation: a Randomized Controlled Exploratory Study (CANVAS-Ⅱ)
Brief Title: Choice of Anesthesia for Endovascular Treatment of Acute Ischemic Stroke in Posterior Circulation
Acronym: CANVAS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-10-15
Record Dates: First submitted 2017-10-15; First posted 2017-10-23 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Posterior Circulation Brain Infarction
Keywords: Anesthesia Methods; Acute Ischemic Stroke; Endovascular Treatment
MeSH Terms: conditions — Brain Infarction; Ischemic Stroke | interventions — Anesthesia, General; Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthesia/conscious sedation (Other): Patients will be injected by propofol (adjusted by bispectral index scale ≥70 ) and /or remifentanil（0.01-0.06μg/kg/min）. Patients will maintain spontaneous breathing.
  Interventions: Procedure: Local anesthesia/concious sedation; Procedure: Spontaneous breath
- General anesthesia (Other): Patients will be induced with remifentanil (0.2-0.8 μg/kg), propofol (1-2mg/kg) and rocuronium (0.6 mg/kg). Anesthesia will then be maintained keep the BIS between 40 and 60 with propofol and remifentanil. After tracheal intubation, patients will be kept with controlled ventilation.
  Interventions: Procedure: General anesthesia; Procedure: Controlled ventilation

INTERVENTIONS:
Procedure: General anesthesia — Patients will be injected with propofol, remifentanil and muscular relaxant with controlled ventilation.
  Arms: General anesthesia
Procedure: Local anesthesia/concious sedation — Patients will be injected with propofol and remifentanil.
  Arms: Local anesthesia/conscious sedation
Procedure: Spontaneous breath — Patients will be kept spontaneous breath.
  Arms: Local anesthesia/conscious sedation
Procedure: Controlled ventilation — Patient will be kept with controlled ventilation.
  Arms: General anesthesia

SUMMARY:
There is few randomized controlled clinical to investigated the impact of anesthetic type on outcome in patients with acute ischemic stroke in posterior cerebral circulation. It is unknown whether the choice of anesthesia is impacted on the outcomes for these patients or not. The investigators will perform a randomized controlled pilot clinical trial of general anesthesia versus local anesthesia/conscious sedation to explore and find out a potential fact whether anesthetic type alters perioperative neurological function in patients with acute ischemic stroke in posterior cerebral circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke in posterior cerebral circulation scheduled to receive emergency endovascular treatment; Age > 18; The onset time is within 24 hours; Modified rankin score ≤2 before onset.

Exclusion Criteria:

* Radiological ambiguity concerning infarction and vessel occlusion; Additional intracerebral hemorrhage; Anterior circulation infraction; Coma on admission (Glasgow coma score less than 8); NIHSS less than 6 or more than 30; Severe agitation or seizures on admission; Obvious loss of airway protective reflexes and/or vomiting on admission; Being intubated before treatment on admission; Known allergy to anesthetic or analgesic;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
modified rankin score（mRS） | post-procedural 90 days
  Modified rankin score（mRS）is used to evaluate the primary outcome. The scale of mRS is 0 to 6. The best neurological outcome is the mRS with 0, indicating no any symptom left, and a good neurological outcome is agreed with a mRS≤2. mRS of 6 is the worst, indicating death. mRS will be evaluated by outcomes assessor who is blinded to the grouping.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Ruquan Han, Fengtai, Beijing Municipality
  - Fan Wang, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang F, Wu Y, Wang X, Yan L, Zhang S, Jian M, Liu H, Wang A, Wang F, Han R; CANVAS II Group. General Anesthesia vs Conscious Sedation for Endovascular Treatment in Patients With Posterior Circulation Acute Ischemic Stroke: An Exploratory Randomized Clinical Trial. JAMA Neurol. 2023 Jan 1;80(1):64-72. doi: 10.1001/jamaneurol.2022.3018. PMID 36156704
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Liang F, Zhao Y, Yan X, Wu Y, Li X, Zhou Y, Jian M, Li S, Miao Z, Han R, Peng Y. Choice of ANaesthesia for EndoVAScular treatment of acute ischaemic stroke at posterior circulation (CANVAS II): protocol for an exploratory randomised controlled study. BMJ Open. 2020 Jul 31;10(7):e036358. doi: 10.1136/bmjopen-2019-036358. PMID 32737091